CLINICAL TRIAL: NCT06764784
Title: The Efficacy of Freehand, Pilot Drilled and Fully Guided Implant Surgery in Partially Edentulous Patients: a Randomize Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Assistant Professor, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECM#2024-3195
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Partial Edentulism Class 1; Dental Implantation; Osseointegration
Keywords: Partial edentulism; Dental implants; Freehand implant surgery; Pilot-drilled implant surgery; Fully guided implant surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Freehand Implant Surgery (Experimental): Participants in this arm will undergo implant placement using the freehand technique. This approach relies on the surgeon's clinical judgment and visual landmarks for implant positioning without the use of specialized guides.
  Interventions: Procedure: Freehand Implant Surgery
- Pilot-Drilled Implant Surgery (Experimental): Participants in this arm will undergo implant placement using the pilot-drilled technique. A pilot drill will be used to create an initial guided pathway for the implant, improving placement accuracy while allowing for some flexibility during the procedure.
  Interventions: Procedure: Fully Guided Implant Surgery
- Fully Guided Implant Surgery (Experimental): Participants in this arm will undergo implant placement using the fully guided technique. This approach utilizes computer-aided surgical templates created from preoperative imaging to ensure precise implant positioning, angulation, and depth
  Interventions: Procedure: Pilot-Drilled Implant Surgery

INTERVENTIONS:
Procedure: Freehand Implant Surgery — This intervention involves implant placement performed manually by the surgeon without the use of specialized guides. The procedure relies on the surgeon's clinical judgment and experience to determine the implant's positioning, angulation, and depth.
  Arms: Freehand Implant Surgery
Procedure: Pilot-Drilled Implant Surgery — This intervention utilizes a pilot drill to create an initial guide hole for the implant. The pilot-drilled pathway improves accuracy while still allowing the surgeon flexibility during the procedure. The final implant is placed following sequential drilling.
  Arms: Fully Guided Implant Surgery
Procedure: Fully Guided Implant Surgery — This intervention employs computer-aided surgical templates created from preoperative imaging data, such as CBCT scans. These guides ensure precise implant positioning, angulation, and depth based on preoperative planning. The approach minimizes variability and enhances accuracy.
  Arms: Pilot-Drilled Implant Surgery

SUMMARY:
This study evaluates three different methods of dental implant surgery-freehand, pilot-drilled, and fully guided techniques-in patients with partial tooth loss (partial edentulism). Dental implants are widely used to restore missing teeth, but the success of these procedures depends heavily on accurate placement and surgical precision.

The study involves 90 participants, divided into three groups of 30, each undergoing one of the three surgical techniques. The main goals are to compare surgery duration, implant placement accuracy, post-operative recovery, patient satisfaction, and long-term success rates.

Key findings suggest that fully guided implant surgery offers the highest accuracy, the shortest recovery time, and the highest patient satisfaction. Pilot-drilled surgery also showed excellent results, providing a balance between precision and efficiency. Freehand surgery, while flexible, showed slightly lower accuracy and higher complication rates.

This research aims to guide patients and healthcare providers in selecting the most suitable implant surgery method for improved outcomes and long-term success in dental care.

DETAILED DESCRIPTION:
This randomized controlled trial will investigate the efficacy of three implant placement techniques-freehand, pilot-drilled, and fully guided-in patients with partial tooth loss. The study will explore critical factors such as surgical precision, patient recovery, implant stability, and overall satisfaction. The objective will be to provide evidence-based guidance for selecting optimal surgical techniques tailored to individual patient needs.

Study Design:

Participants: 90 partially edentulous patients will be randomly assigned into three groups (30 patients per group).

Techniques:

Freehand surgery: Surgeons will rely on their skill and judgment for implant placement without specialized guides.

Pilot-drilled surgery: Surgeons will use a pilot drill to create an initial guided pathway for implant placement.

Fully guided surgery: Computer-aided templates will be utilized for precise positioning based on preoperative imaging and planning.

Outcomes Measured:

Surgical Parameters:

Duration of surgery. Intraoperative complications.

Postoperative Recovery:

Pain, swelling, and healing responses.

Implant Stability and Osseointegration:

Radiographic imaging and resonance frequency analysis will assess outcomes at 3, 6, and 12 months.

Patient Satisfaction:

Surveys will measure aesthetics, comfort, and satisfaction with treatment outcomes.

Long-term Success Rates:

Implant survival rates and peri-implant bone health will be evaluated.

Key Findings:

Fully guided surgery is expected to demonstrate superior accuracy, reduced recovery times, and the highest patient satisfaction.

Pilot-drilled surgery is anticipated to offer a robust balance of precision and efficiency, with high implant survival rates.

Freehand surgery may show slightly lower success rates and higher variability in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years.
* Patients with partial edentulism (missing one or more teeth in an otherwise dentate arch).
* Sufficient bone volume and quality to support implant placement without additional bone augmentation.
* Good overall health with no systemic contraindications for surgery.
* Willingness to provide informed consent and comply with the study protocol and follow-up visits.

Exclusion Criteria:

* Patients with uncontrolled systemic conditions (e.g., diabetes, cardiovascular diseases) that may affect healing or surgery outcomes.
* Pregnant or lactating women.
* Smokers or individuals with a history of poor compliance with post-operative care.
* Patients requiring additional bone grafting, sinus lifts, or complex augmentation procedures for implant placement.
* Active oral infections, untreated periodontal disease, or severe malocclusion that could interfere with implant placement or outcomes.
* Patients with a history of bisphosphonate use or other medications known to affect bone metabolism.
* Individuals with mental or physical conditions that would impair their ability to participate in the study or follow the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of Implant Placement | Immediately post-surgery
  Accuracy of implant positioning will be assessed using postoperative radiographic imaging (CBCT) to measure deviations in angulation, depth, and position from the preoperative plan.
Postoperative Complication | Within 2 weeks post-surgery
  Incidence of complications such as bleeding, infection, nerve damage, or soft tissue trauma will be recorded.

SECONDARY OUTCOMES:
Surgery Duration | During the surgical procedure
  The time required for implant placement will be measured from the start of the surgery to the placement of the implant.
Pain Levels | Days 1, 3, and 7 post-surgery
  Pain will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain).
Implant Stability | At 3, 6, and 12 months post-surgery
  Resonance frequency analysis (RFA) will be used to measure the implant stability quotient (ISQ).

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns related to patient privacy and confidentiality. Although the study will follow rigorous data collection and management protocols, sharing raw participant data might compromise the anonymity and security of the participants' health information. Additionally, the data may be specific to the study design and not directly generalizable, limiting its applicability to external research.